CLINICAL TRIAL: NCT06847165
Title: Trigeminal Nerve Stimulation for Children With Prenatal Alcohol Exposure
Acronym: TNS-PAE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Joseph O'Neill, PhD, Professor of Child Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-0648; R61AA031029 (NIH)
Record Dates: First submitted 2025-02-16; First posted 2025-02-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Fetal Alcohol Spectrum Disorders; Attention Deficit Hyperactivity Disorder
Keywords: prenatal alcohol exposure; attention deficit hyperactivity disorder; trigeminal nerve stimulation
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: open label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Trigeminal Nerve Stimulation (Experimental): Each child will receive nightly trigeminal nerve stimulation, administered by the parent at bedtime, for 8 hrs while sleeping overnight, nightly for 4 weeks (28 days)
  Interventions: Device: Trigeminal Nerve Stimulation (TNS)

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation (TNS) — In TNS, a weak electric current is applied to the child's forehead overnight while sleeping to gently stimulate the brain. TNS treatment is typically administered at home at bedtime by the parent to the child. The TNS device is small (size of a cell phone) and easy to use. Two thin wires go from the device to a pair of small electrodes that tape onto the forehead like a band-aid. The parent presses three keys on the device and it is ready to go.
  Other Names: external trigeminal nerve stimulation

SUMMARY:
This is an open-label trial of trigeminal nerve stimulation (TNS) for children aged 8-12 years with attention deficit hyperactivity disorder (ADHD) putatively due to prenatal alcohol exposure (PAE). TNS has been successful in treating pediatric ADHD generally and it is US Food and Drug Administration (FDA)-cleared for this condition. But this will be the first time it is tried for ADHD specifically associated with PAE. In TNS, a weak electric current is applied to the child's forehead overnight while sleeping to gently stimulate the brain. TNS is administered at home by the parent to the child. TNS is safe and well tolerated. Efficacy of TNS in ADHD is ~50%. The purpose of the present pilot study is to determine the feasibility of TNS for children with PAE and ADHD. Feasibility means safety (any serious side effects?), tolerability (do children comply with TNS? are they comfortable with it?), and a rough idea of efficacy (does TNS seem to work in most kids?) A secondary goal of the study is to get a more precise idea of brain mechanisms of TNS with magnetic resonance imaging (MRI). Families who participate will make three clinic visits: eligibility (4-5 hours), pre-TNS (2-3 hours including MRI), and post-TNS (2-3 hours including MRI). Children will receive TNS, applied by the parent, for 8 hours every night while sleeping for 4 weeks. Four weeks after treatment, families will take part in a telephone follow-up, to see whether any improvements made last.

DETAILED DESCRIPTION:
Trigeminal nerve stimulation (TNS) is a new treatment for pediatric ADHD developed at University of California Los Angeles (UCLA). In TNS, a weak electric current is applied to the child's forehead overnight while sleeping to gently stimulate the brain. TNS treatment is typically administered at home at bedtime by the parent to the child. The TNS device is small (size of a cell phone) and easy to use. Two thin wires go from the device to a pair of small electrodes that tape onto the forehead like a band-aid. The parent presses three keys on the device and it is ready to go. TNS is safe and well tolerated. The success rate, or efficacy, of TNS is about 50% in children with ADHD overall. Although TNS is FDA-cleared for children with ADHD, regardless of the cause, or etiology, of the ADHD, the possible influence of etiology on TNS success has not yet been studied. One common etiology of ADHD is prenatal alcohol exposure (PAE). When a mother drinks alcohol during pregnancy her child often develops ADHD. While TNS is an approved treatment for these children, it is actually not known whether they would respond any differently. It is known that drug treatments that routinely work well in children with ADHD without PAE are poorly effective in many children with ADHD due to PAE. Thus, there is a chance children with ADHD due to PAE could respond differently (better or worse) to TNS as well. The purpose of the research is to determine the safety and efficacy of TNS specifically in children whose ADHD is associated with PAE. We expect that TNS will be as safe and effective in children with ADHD with PAE as in children without, but that needs to be formally tested. As a first step in the formal testing process, this pilot study aims to determine the feasibility of TNS in children with ADHD associated with PAE. Feasibility means safety (any serious side effects?), tolerability (do children comply with TNS? are they comfortable with it?), and a rough idea of efficacy (does TNS seem to work in most kids?) A secondary goal of our study is to get a more precise idea of where and how TNS acts in the brain using MRI-based neuroimaging. Families who participate in the study will come to the clinic for three visits: eligibility (4-5 hours), pre-TNS (2-3 hours including MRI), and post-TNS (2-3 hours including MRI). Thus, the child will undergo two MRIs of the brain, a safe, non-invasive, and radiation-free procedure. The child will receive TNS treatment, applied by the parent, for 8 hours every night while sleeping for 4 weeks. Four weeks after treatment, families will take part in a telephone follow-up, to see whether any improvements made last.

ELIGIBILITY:
Inclusion Criteria:

* - Fetal alcohol syndrome, partial fetal alcohol syndrome, or alcohol-related neurodevelopmental disorder per modified Institute of Medicine criteria (thus positive maternal drinking in pregnancy required, facial stigmata not required)
* Prenatal alcohol exposure (PAE) >6 drinks/week for >= 2 weeks and/or >= 3 drinks on >= 2 occasions throughout gestation per Health Interview for Women/Health Interview for Adoptive and Foster Parents (HIW/HIAFP)
* Diagnosis of Diagnostic and Statistical Manual 5th edition (DSM-5) attention deficit hyperactivity disorder (ADHD), including problems with inattention, hyperactivity, impulsivity, and/or executive function. Screening for ADHD will be done using the Swanson, Nolan, and Pelham Teacher and Parent Rating Scale (SNAP IV). Formal diagnosis of ADHD will be based on the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) with input from the Behavior Rating of Executive Function (BRIEF II) and the Conners 4.
* Parent and child able to complete testing in English
* Child able to cooperate during MRI
* Full-Scale Intelligence Quotient >70 per the Kaufman Brief Intelligence Test (K-BIT-2)
* Child able to comply with study procedures
* Age 8-12

Exclusion Criteria:

* - Other toxic exposure per HIW/HIAFP whose influence clearly surpasses that of alcohol (very rare) per study clinician judgement
* Known genetic syndrome associated with ADHD-like symptoms including fragile X, tuberous sclerosis, or generalized resistance to thyroid hormone
* Serious medical or neurologic illness likely to influence brain function, e.g., seizures, closed-head trauma
* Gestation < 34 weeks
* Ferromagnetic metal, claustrophobia, or other MRI or TNS contraindication (e.g., insulin pumps or other body-worn devices)
* Diagnosis of autism spectrum disorder, psychotic disorder, or major mood disorder
* Active suicidal ideation as evidenced by meeting criteria for "Current" or "Lifetime attempt" on the Suicidality module or "Current' or 'In early remission' on the Suicide Behavior Disorder module of the MINI KID

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-04-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale Total Score | administered at baseline and up to 1 week after completing 4 weeks of trigeminal nerve stimulation (TNS) treatment
  clinician-administered measure of severity of core ADHD symptoms: inattention and hyperactivity/impulsivity; minimum score 0, maximum score 40, a higher score means a worse outcome

SECONDARY OUTCOMES:
Clinical Global Impression-- Severity (CGI-S) for Attention Deficit Hyperactivity Disorder (ADHD) | administered at baseline
  This is clinician-administered measure of overall severity of ADHD symptoms: minimum score 1, maximum score 7; higher score is worse outcome
Clinical Global Impression-- Improvement (CGI-I) for ADHD | administered up to 1 week after completing 4 weeks of trigeminal nerve stimulation (TNS) treatment
  CGI-I: minimum score 1, maximum score 7; higher score is worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Joseph O'Neill, PhD, Principal Investigator — UCLA Division of Child & Adolescent Psychiatry
Locations (1):
- University of California Los Angeles Semel Institute Division of Child & Adolescent Psychiatry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be posted to the National Institute on Alcohol Abuse and Alcoholism (NIAAA) Data Archive
Time Frame: Data posted to the NIAAA Data Archive will be updated every 6 months after enrollment of the first subject. Data will remain posted in perpetuity or until the Archive takes them down.
Access Criteria: Any investigator with access to the NIAAA Data Archive will have access to the data.
URL: https://www.niaaa.nih.gov/research/data-archive-and-resources/niaaa-data-archive

REFERENCES:
- [Derived] O'Neill J, Joshi S, Alger JR, Leuchter AF, Schneider BN, O'Connor MJ. Trigeminal nerve stimulation (TNS) for children with attention deficit/hyperactivity disorder and fetal alcohol spectrum disorder: Feasibility study protocol. PLoS One. 2025 Aug 29;20(8):e0330986. doi: 10.1371/journal.pone.0330986. eCollection 2025. PMID 40880352
- [Derived] O'Neill J, Joshi S, Alger JR, Schneider BN, O'Connor MJ. Trigeminal Nerve Stimulation (TNS) for Children with Attention Deficit/Hyperactivity Disorder and Fetal Alcohol Spectrum Disorder: Feasibility Study Protocol. medRxiv [Preprint]. 2025 Jul 7:2025.07.07.25331025. doi: 10.1101/2025.07.07.25331025. PMID 40672490